CLINICAL TRIAL: NCT04161560
Title: Cetuximab - IRDye800 Intraoperative Fluorescence Imaging in Esophagectomy of Esophageal Cancer:A Single Center Clinical Research
Brief Title: Cetuximab - IRDye800 Intraoperative Fluorescence Imaging in Esophagectomy of Esophageal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MIC-ESO-001
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Drug Safety ; Drug Specificity
Keywords: Cetuximab-IRDye800; EGFR; esophageal squamous cell carcinoma; real-time imaging
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Intervention Model Description: 1， dose of drug 2, control group
Masking Description: 4 groups according to different doses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- use of the cetuximab-IRDye800 (Experimental): four groups : control group, 1% dose group (1% of therapeutic dose; 2.5 Mg/m2) and 10% dose groups (10%of therapeutic dose ;25mg/m2) and 25% dose group (25%of therapeutic dose; 62.5mg/m2)
  Interventions: Drug: Cetuximab-IRDye800

INTERVENTIONS:
Drug: Cetuximab-IRDye800 — does of Cetuximab-IRDye800

SUMMARY:
The esophageal squamous cell carcinoma (ESCC) has high prevalence and mortality in China, which become a severe challenge for public health. The molecular imaging technology has been developed for intra-operative visualization and precise resection of the tumors. The imaging probe possess high affinity to the tumor specific targets. Among the tumor related proteins, EGFR is located on the cell membrane and over expresses in more than 50% ESCC which has been used as an ideal target for molecular imaging.

Cetuximab is an EGFR targeting antibody for anti cancer therapy. When labeled with an commercial available fluorescence dye IRDye800, cetuximab has been used as molecular imaging probe in clinical trials for surgical navigation of cancers including head and neck squamous cell cancers and gliomas. Previous studies shown high safety when using this probe and excellence sensitivity for cancer detection, which bring great promise in translational medicine.

This is a single-center prospective sequential trial. It is the first attempt to apply cetuximab-IRDye800 probe in ESCC surgery. This probe will be produced under clinical Good Manufacturing Practice (cGMP) conditions. The ESCC patients will be recruited with strict criteria.Patients population is planned to be 40 cases between18 and 65 years old, without gender limit. The patients will be divided into four groups : control group without probe administration, 1% dose group (1% of therapeutic cetuximab dose; 2.5 Mg/m2) and 10% dose groups (10%of therapeutic cetuximab dose ;25mg/m2) and 25% dose group (25%of therapeutic cetuximab dose; 62.5mg/m2), 10 cases are sequential assigned to each group. After informed consent, patients will receive a systemic infusion of the study drug 2 days before surgery.

Primary (safety and efficiency) and secondary endpoints (tissue EGFR expression) will be recorded. Preoperative management and surgical procedures will been performed according to conventional protocols. Intra-operative imaging of the surgical field will be performed in real time at 2 time points: before and post tumor resection. The postoperative specimens will be subjected to pathological analysis including correlation study of fluorescence signal and tumor tissue in pathology slice.

A protocol for managing any allergic reaction related to systemic infusion of cetuximab has been established. The patient's vital signs and ECG will be closely monitored post probe administration. The blood, liver and kidney, coagulation function and cardiotoxicity will be evaluated before and post surgery.

This clinical trial is anticipated to validate the concept that intra-operative fluorescent imaging of esophageal squamous cell carcinoma with cetuximab-IRDye800 can facilitate the demarcation of tumor boundary and identification of metastatic lymph nodes and testify its safety.

ELIGIBILITY:
Inclusion Criteria:

1.18 years old ≤ age ≤ 65 years old, gender is not limited; 2. Esophageal squamous cell carcinoma confirmed by cytology or histology and requiring surgical treatment; 3. Preoperative high-grade gastroscopy confirmed that the tumor staging was T1-3N0-1M0 patients feasible for surgical resection; 4. The main organ function is basically normal: Karnofsky score >70%; 5. Laboratory blood tests meet surgical safety standards; 6. Informed consent form is signed before the study, the patient and / or their legal representative have the ability to fully understand the content of the trial, the process and possible adverse reactions, and the patients are able to comply for regular visit; 7. Women of reproductive age must have a negative pregnancy test and are not breastfeeding, both men and women need to receive contraceptive methods approved by the investigator and agree to maintain this contraceptive from the date of signing the informed consent to the end of the study.

Exclusion Criteria:

1. Cetuximab drug allergy sufferers;
2. Preoperative electrocardiogram indicates patients with prolonged QTc interval;
3. People with mental or neurological diseases;
4. Patients with cachexia and severe malnutrition;
5. Patients with surgical contraindications such as coagulopathy, HIV antibody positive, and severely poorly controlled clinical infections;
6. Patients with other combined diseases (such as abnormal liver and kidney function) or combined medications, which may be affected by the investigator.
7. Patients who are simultaneously involved in another clinical study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Tumor to Background Ratio | intra-operative
  Tumor to Background Ratio by mean fluorescence intensity in tumor tissue and lymph nodes
relative adverse drug reaction | 14 days after using cetuximab-IRDye800
  relative adverse drug reaction after using cetuximab-IRDye800

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miller SE, Tummers WS, Teraphongphom N, van den Berg NS, Hasan A, Ertsey RD, Nagpal S, Recht LD, Plowey ED, Vogel H, Harsh GR, Grant GA, Li GH, Rosenthal EL. First-in-human intraoperative near-infrared fluorescence imaging of glioblastoma using cetuximab-IRDye800. J Neurooncol. 2018 Aug;139(1):135-143. doi: 10.1007/s11060-018-2854-0. Epub 2018 Apr 6. PMID 29623552
- [Result] Rosenthal EL, Moore LS, Tipirneni K, de Boer E, Stevens TM, Hartman YE, Carroll WR, Zinn KR, Warram JM. Sensitivity and Specificity of Cetuximab-IRDye800CW to Identify Regional Metastatic Disease in Head and Neck Cancer. Clin Cancer Res. 2017 Aug 15;23(16):4744-4752. doi: 10.1158/1078-0432.CCR-16-2968. Epub 2017 Apr 26. PMID 28446503
- [Result] Rosenthal EL, Warram JM, de Boer E, Chung TK, Korb ML, Brandwein-Gensler M, Strong TV, Schmalbach CE, Morlandt AB, Agarwal G, Hartman YE, Carroll WR, Richman JS, Clemons LK, Nabell LM, Zinn KR. Safety and Tumor Specificity of Cetuximab-IRDye800 for Surgical Navigation in Head and Neck Cancer. Clin Cancer Res. 2015 Aug 15;21(16):3658-66. doi: 10.1158/1078-0432.CCR-14-3284. Epub 2015 Apr 22. PMID 25904751
- [Result] Korb ML, Hartman YE, Kovar J, Zinn KR, Bland KI, Rosenthal EL. Use of monoclonal antibody-IRDye800CW bioconjugates in the resection of breast cancer. J Surg Res. 2014 May 1;188(1):119-28. doi: 10.1016/j.jss.2013.11.1089. Epub 2013 Nov 22. PMID 24360117
- [Result] Sturm MB, Joshi BP, Lu S, Piraka C, Khondee S, Elmunzer BJ, Kwon RS, Beer DG, Appelman HD, Turgeon DK, Wang TD. Targeted imaging of esophageal neoplasia with a fluorescently labeled peptide: first-in-human results. Sci Transl Med. 2013 May 8;5(184):184ra61. doi: 10.1126/scitranslmed.3004733. PMID 23658246
- [Result] van Dam GM, Themelis G, Crane LM, Harlaar NJ, Pleijhuis RG, Kelder W, Sarantopoulos A, de Jong JS, Arts HJ, van der Zee AG, Bart J, Low PS, Ntziachristos V. Intraoperative tumor-specific fluorescence imaging in ovarian cancer by folate receptor-alpha targeting: first in-human results. Nat Med. 2011 Sep 18;17(10):1315-9. doi: 10.1038/nm.2472. PMID 21926976
- [Result] Bird-Lieberman EL, Neves AA, Lao-Sirieix P, O'Donovan M, Novelli M, Lovat LB, Eng WS, Mahal LK, Brindle KM, Fitzgerald RC. Molecular imaging using fluorescent lectins permits rapid endoscopic identification of dysplasia in Barrett's esophagus. Nat Med. 2012 Jan 15;18(2):315-21. doi: 10.1038/nm.2616. PMID 22245781
- [Result] Petty RD, Dahle-Smith A, Stevenson DAJ, Osborne A, Massie D, Clark C, Murray GI, Dutton SJ, Roberts C, Chong IY, Mansoor W, Thompson J, Harrison M, Chatterjee A, Falk SJ, Elyan S, Garcia-Alonso A, Fyfe DW, Wadsley J, Chau I, Ferry DR, Miedzybrodzka Z. Gefitinib and EGFR Gene Copy Number Aberrations in Esophageal Cancer. J Clin Oncol. 2017 Jul 10;35(20):2279-2287. doi: 10.1200/JCO.2016.70.3934. Epub 2017 May 24. PMID 28537764
- [Result] Hu XY, Wang R, Jin J, Liu XJ, Cui AL, Sun LQ, Li YP, Li Y, Wang YC, Zhen YS, Miao QF, Li ZR. An EGFR-targeting antibody-drug conjugate LR004-VC-MMAE: potential in esophageal squamous cell carcinoma and other malignancies. Mol Oncol. 2019 Feb;13(2):246-263. doi: 10.1002/1878-0261.12400. Epub 2018 Nov 15. PMID 30372581